CLINICAL TRIAL: NCT06189222
Title: The Effect of Virtual Reality Glasses Used During Intravenous Catheter Insertion on The Child's Emotional Responses
Brief Title: The Effect of Virtual Reality Glasses Used During Intravenous Catheter Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Türkan Şen (Other)
Responsible Party: Sponsor-Investigator, Türkan Şen, Professional Nurse, Pamukkale University
Organization: Pamukkale University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PamukkaleU-SBF-TŞ-01
Record Dates: First submitted 2023-12-07; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Anxiety and Fear
Keywords: Invasive procedures, Pediatrics, Emotion, Fear, Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: study group: children evaluated with virtual reality glasses control group: children receiving standard care
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality glasses (Experimental): The sample of the research, which was carried out as a randomized controlled experimental study, consisted of 102 children, including 51 in the control group and 51 in the study group, who were aged between 7 and 12 and were on treatment in the emergency department. Research data were collected using a Descriptive Data Form for Children and the Children's Emotional Manifestation Scale. During the data collection phase, first, the Descriptive Data Form for Children was filled out for the control and study groups. No intervention was applied to the control group. After the tourniquet was tied in the study group, the children started watching a video of their choice through virtual reality glasses. When the process was completed, the video was stopped. During this period, the child was evaluated using the Children's Emotional Manifestation Scale.
  Interventions: Device: virtual reality glasses
- standard care (No Intervention): Intervention during intravenous catheter insertion to the child

INTERVENTIONS:
Device: virtual reality glasses — The population of the study consisted of children who were aged between 7- 12 and were on treatment using an intravenous catheter in the pediatric emergency unit of a state hospital in Turkey.Participants were divided into two groups, namely experimental and control groups, by using simple randomization software. The design and implementation of the study were based on the principles in the CONSORT list (Consolidated Standards of Reporting Studies). Descriptive data form for children,this form was prepared to collect information about the children included in the sample. It consists of seven questions on children's sociodemographic characteristics and previous intravenous catheter insertion experience.The Children's Emotional Manifestation Scale (CEMS), this scale was developed by Li & Lopez (2005) to measure children's emotional responses during stressful medical procedures. The VR glasses we used in our study were connected to a mobile phone.
  Arms: virtual reality glasses

SUMMARY:
The purpose of this clinical trial is to evaluate the effect of the virtual reality glasses device on the child's emotional responses during invasive interventions in child health services.

The main question it aims to answer are:

- Is there a difference between the emotional responses of children who watched cartoons with virtual reality glasses (experimental group) and the children in the control group during the intravenous catheter insertion process? First, the descriptive data form for the children was filled out for the control and study groups. Then, to distract the children during the application of the intravenous catheter, they watched cartoon videos of their choice for the 7-12 age group through virtual reality glasses by using a free internet application throughout the procedure. The procedure started with tying the tourniquet and continued until the intravenous catheter insertion was completed. During this period, the child's emotional responses were evaluated with the Children's Emotional Manifestation Scale. No intervention was applied to the control group. throughout the process the child's emotional responses were evaluated with the Children's Emotional Manifestation Scale.

No intervention was applied to the control group.

DETAILED DESCRIPTION:
This study was conducted to determine the effect of virtual reality glasses used during intravenous catheter insertion on the child's emotional responses. The sample of the research, which was carried out as a randomized controlled experimental study, consisted of 102 children, including 51 in the control group and 51 in the study group, who were aged between 7 and 12 and were on treatment in the emergency department. Research data were collected using a Descriptive Data Form for Children and the Children's Emotional Manifestation Scale. During the data collection phase, first, the Descriptive Data Form for Children was filled out for the control and study groups. No intervention was applied to the control group. After the tourniquet was tied in the study group, the children started watching a video of their choice through virtual reality glasses. When the process was completed, the video was stopped. During this period, the child was evaluated using the Children's Emotional Manifestation Scale. A statistically significant difference was found between the Children's Emotional Manifestation Scale scores of the children in the study and control groups. The scores of the children in the study group were statistically significantly lower than the scores of the children in the control group.During the intravenous catheter insertion process, children who watched cartoons on virtual reality glasses showed less negative emotional behavior than those who did not.The use of virtual reality glasses is a developing technology in child health services, and it is recommended to encourage their use in these services.

ELIGIBILITY:
Inclusion Criteria:

* Children who

  * were aged 7-12,
  * had parental permission,
  * gave verbal consent,
  * and whose parents could speak Turkish,
  * were conscious,
  * and did not have orthopedic, neurological, or sight-related problems that prevented wearing virtual reality glasses were included in the study.

Exclusion Criteria:

* Children who

  * had a chronic disease that required frequent vascular access,
  * had visual and hearing impairments,
  * had a mental and neurological disability,
  * had previously participated in a similar study,
  * had a febrile illness at the time of application,
  * had a history of fainting during vascular access procedures, or
  * had used medication in the last 24 hours before the application, which might have an analgesic effect, were not included in the study.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
The Children's Emotional Manifestation Scale (CEMS) | 7 months
  The scale, which allows direct behavioral observation, consists of five different behavioral categories, namely facial expression, vocalization, activity, interaction, and level of cooperation. Each category includes five different observable behaviors rated by level and intensity. The scale is scored by reviewing descriptions of the behavior in each category and selecting the value that most represents the observed behavior. Each category is scored from 1 to 5. The scores obtained for each category are summed and a total score between 5- 25 is obtained. High scale scores indicate the exhibition of more negative emotional behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)